CLINICAL TRIAL: NCT07014059
Title: "In Vivo Evaluation of Topical Ocular Use of Autologous Serum Obtained by a Closed-Circuit Collection Device."
Brief Title: Autologous Serum Obtained by a Closed-Circuit Collection Device
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GIANCARLO FATOBENE (Other)
Collaborators: JP Farma (Unknown)
Responsible Party: Sponsor-Investigator, GIANCARLO FATOBENE, MD, PhD, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 78127624.4.0000.0068
Record Dates: First submitted 2025-01-21; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: GVHD; Meibomian Gland Dysfunction (Disorder); Stevens-Johnson Syndrome; Limbal Keratoconjunctivitis; Recurrent Erosions of Persistent Epithelial Defects; Neurotrophic Ulcer; Sjogren Syndrome With Keratoconjunctivitis
Keywords: soro autologo; gvhd; Sjogren's Syndrome (SS); Meibomian Gland Dysfunction (Disorder); Stevens-Johnson Syndrome; Limbal Keratoconjunctivitis; Neurotrophic Ulcer; Recurrent Erosions of Persistent Epithelial Defects; Study Protocol - Autologous Serum; Autologous Serum
MeSH Terms: conditions — Meibomian Gland Dysfunction; Stevens-Johnson Syndrome; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Production of autologous serum in a closed system for ocular use (Experimental)
  Interventions: Drug: Autologous Serum 20%

INTERVENTIONS:
Drug: Autologous Serum 20% — The collection of autologous serum in a closed blood processing system for ocular use

SUMMARY:
Autologous serum eye drops (ASED) are an established therapy for ocular surface diseases; however, their preparation can be costly and may not be available due to the need for germ-free conditions. This pilot trial assesses the feasibility of collecting ASED in a closed-circuit system for patients with chronic ocular surface diseases.

DETAILED DESCRIPTION:
Autologous Serum exhibits characteristics very similar to those of tears, such as pH, osmolarity, vitamins, and Immunoglobulin A. It also contains growth factors, nutritional factors, and antibacterial components that are necessary for the maintenance of cellular viability in the epithelial repair process. The use of autologous serum eye drops was first described in 1984 by Fox et al., in research for a preservative-free tear substitute. Subsequently, in 1999, Tsubota et al. found that, due to the presence of growth factors and vitamins, autologous serum could have a true epithelial trophic potential for the ocular surface. The autologous serum eye drops are not only a lubricant for the ocular surface but also provide various essential substances for the reconstruction of epithelial damage, including vitamin A, epithelial growth factor, fibronectin, and a variety of cytokines. With these epithelial trophic factors, autologous serum facilitates proliferation, migration, and differentiation of the ocular surface epithelium. Moreover, it is known for its anti-catabolic properties, inhibiting the inflammatory cascade triggered by interleukin-1, which prevents tissue destruction. Therefore, autologous serum eye drops have been effective in the treatment of persistent epithelial defects, neurotrophic ulcers, superior limbic keratoconjunctivitis, dry eye conditions, graft-versus-host disease (GVHD), or after refractive surgeries, such as LASIK (Laser Assisted In Situ Keratomileusis). In 2020, Wang et al. published an article with 7 randomized controlled trials comparing the use of autologous serum versus artificial tears in patients with dry eye syndrome. In the meta-analysis, all 7 studies evaluated subjective symptoms and showed that autologous serum eye drops were superior to ocular lubricants in alleviating and remitting symptoms. It was shown that autologous serum eye drops significantly improved parameters such as OSDI (Ocular Surface Disease Index), tear break-up time, and Bengal Rose staining when compared to the control group using ocular lubricants. Given the numerous properties of autologous serum eye drops, there is no doubt about their benefit and effectiveness in treating several ocular surface diseases, including ocular GVHD. However, the difficulty in accessing production and the substantial cost of autologous serum eye drops are the main challenges, and their use is often limited to more severe dry eye cases and those refractory to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Dry eye and/or chronic epithelial defects of the ocular surface with indication for autologous serum according to the evaluation of ophthalmologists specialized in Cornea and Ocular Surface;
* Peripheral venous access or PICC that allows the collection of whole blood.

Exclusion Criteria:

* Active ocular infection;
* Hemoglobin < 11 g/dL;
* Angina, MI, or stroke in the last 30 days;
* Significant pulmonary or cardiac disease that contraindicates autologous serum collection in the investigator's opinion;
* Active ocular or systemic infection at the time of collection;
* Inability to attend follow-up visits at 6 and 12 weeks;
* Active hematological malignancy (except measurable residual disease) or solid malignancy (except non-melanoma skin cancer);
* Positive for HIV, HCV, HBV, HTLV, Chagas disease, or syphilis;
* Life expectancy < 6 months;
* Not pregnant (as reported by the participant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using the collection device under testing | 2 years
  Proportion of blood collections that resulted in successful production of final autologous serum containers suitable for patient use.

SECONDARY OUTCOMES:
Median pre-freezing number of leukocytes in autologous serum | 2 years
  0.0-0.03x10ˆ3/mcL;
Median pre-freezing number of red blood cells in autologous serum | 2 years
  0.0-0.03x10ˆ6/mcL;
Median pre-freezing number of platelets in autologous serum | 2 years
  0.0-0.03x10ˆ3/mcL;
Median pre and post-freezing pH in autologous serum | 2 years
  7.00-7.50;
Pre-freezing microbiological test of autologous serum | 2 years
  Positive or negative;
NIH ocular score | baseline, 6 weeks, 12 weeks, and end of treatment
  0-3
Ocular Surface Disease Index | Baseline, 6 weeks, 12 weeks, and end of treatment
  Reported by the patient from 0 to 100
Global ocular symptom score | Baseline, 6 weeks, 12 weeks, and end of treatment
  Reported by the patient from 0 to 10
Lee score ocular subscale | Baseline, 6 weeks, 12 weeks, and end of treatment
  Reported by the patient from 0 to 100
Corneal staining score (fluorescein) | Baseline, 6 weeks, 12 weeks
  Bijsterveld scale: 0-9.
Corneal staining score (Rose Bengal) | Baseline, 6 weeks, 12 weeks
  Bijsterveld scale: 0-9.
Meibography | Baseline, 6 weeks, 12 weeks
  Good, moderate, poor
Schirmer test | Baseline, 6 weeks, 12 weeks
  0-30 mm in 5 minutes
Non-invasive tear film break-up | Baseline, 6 weeks, 12 weeks
  0-50 seconds
Tear film lipid layer | Baseline, 6 weeks, 12 weeks
  0-3
Adherence to the use of autologous serum | At 6 and 12 weeks post-treatment
  Percentage of doses administered vs. planned doses: 0-100%
Patient's qualitative evaluation of the use of autologous serum | At 12 weeks post-treatment
  Qualitative questionnaire
Team's qualitative perception of the feasibility of collection and production of autologous serum | At 50% of planned recruitment
  Qualitative questionnaire

OTHER OUTCOMES:
Pre- and post-growth factor in autologous serum | two years
  EGF, PDGF, NGF, Substance P, hialuronic acida, vitamin A and Vitamin D

CONTACTS AND LOCATIONS:
Locations (1):
- HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided